CLINICAL TRIAL: NCT02834195
Title: Validation of a Classification of Types of Upper Limb and Hand in Patients With Cerebral Palsy
Brief Title: Types of Upper Limb and Hand in Patients With Cerebral Palsy
Acronym: CLASS-MS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D21882
Record Dates: First submitted 2016-07-04; First posted 2016-07-15 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-06

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; reliability; upper limb and hand patterns; classification
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Cerebral palsy (CP) has been defined as "a group of permanent disorders of the development of movement and posture causing activity limitation(s) that are attributed to non-progressive disturbances that occurred in the developing fetal or infant brain".

Investigators previously developed two classification systems, one for the upper limb and one for the hand, based on 100 films of patients with cerebral palsy. Separate classifications were developed following an initial study in which investigators found no correlations between upper limb and hand patterns, meaning that specific upper limb patterns are not always associated with specific hand patterns. Thumb patterns were not included in these classifications since robust classifications already exist, moreover thumb patterns are independent from hand patterns.

The aim is to evaluate the inter- and intra-rater reliability of two previously developed classifications of upper limb and hand patterns.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy

Exclusion Criteria:

* none

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in upper limb pattern classification of each examiner between day 1 and month 2 | examiner classification at day 1 and at month 2.
  Intra-rater reliability of a classification of upper limb pattern in patients with cerebral palsy.
Change in hand pattern classification of each examiner between day 1 and month 2 | examiner classification at day 1 and at month 2.
  Intra-rater reliability of a classification of hand pattern in patients with cerebral palsy.
Change between examiner classification and the expert examiner classification | Expert examiner classification (day 1) and examiner classification (week 4)
  Level of agreement will be determined with Fleiss's kappa (k) and its 95% confidence interval Inter-rater reliability of a classification of upper limb pattern in patients with cerebral palsy.
Change between examiner classification and the expert examiner classification | Expert examiner classification (day 1) and examiner classification (week 4)
  Level of agreement will be determined with Fleiss's kappa (k) and its 95% confidence interval.
  Inter-rater reliability of a classification of hand pattern in patients with cerebral palsy.

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine TOUZET, MD, Principal Investigator — Hospices Civils de Lyon, Pôle Information Médicale, Evaluation, Recherche
Locations (1):
- Hospices Civils de Lyon, Pôle Information Médicale, Evaluation, Recherche - 162 avenue Lacassagne - Bâtiment A, Lyon, France